CLINICAL TRIAL: NCT04257552
Title: Care After Pregnancy Study (CAPS): Randomized Controlled Trial of Patient Engagement After Pregnancy
Brief Title: Care After Pregnancy Study (CAPS): Engaging Women in Postpartum Care
Acronym: CAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Katherine Himes, Associate Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY19040312; 1R56NR017933-01A1 (NIH)
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Results first posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-09

CONDITIONS: Postpartum Care
Keywords: contraception; postpartum care; breast feeding; interconception care
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigators are unaware of study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Attention Control Group (Active Comparator): If randomized to the attention control arm participants will receive discharge instruction from the postpartum nurses per usual care. Study investigators will ask them to provide us with an SMS number. This will enable collection of self-reported breast feeding duration as well as texts on general infant care. The infant care texts are educational in nature and no data will be collected. Participants will receive a total of two texts on general infant care in the first month postpartum. This increased attention to the control arm mirrors the attention received by the Healthy Beyond Pregnancy arms and seeks to isolate the effect of the intervention from a general increased level of contact with providers.
  Interventions: Other: Attention Control
- Pre-Scheduled Postpartum Visit: (Active Comparator): If randomized the usual care with pre-scheduled visit arm, participants will schedule their postpartum visit with the study coordinator and receive discharge information per usual care.
  Interventions: Behavioral: Pre-Scheduled Postpartum Visit
- Healthy Beyond Pregnancy (Experimental): Healthy Beyond Pregnancy is a web platform with an electronic survey that assesses a participant's self-identified postpartum concerns. Participants are then presented with 3 educational videos that reflect their self-identified needs from the survey. The Healthy Beyond Pregnancy generates an individualized passport for postpartum care. This passport for care lists the women's self-identified postpartum needs as well as issues that should be prioritized based on her health history. The individualized passport for postpartum care will be printed out and given to participants. After the participant schedules her postpartum visit, she will receive a printout that includes the date and time of her appointment, a copy of the commitment statement.
  Interventions: Behavioral: Healthy Beyond Pregnancy

INTERVENTIONS:
Behavioral: Healthy Beyond Pregnancy — Web-based application grounded in tenants of behavioral economics.
  Arms: Healthy Beyond Pregnancy
Behavioral: Pre-Scheduled Postpartum Visit — Participants will have their postpartum visit scheduled while they are still in the hospital after delivery.
  Arms: Pre-Scheduled Postpartum Visit:
Other: Attention Control — Participants will receive texts related to infant care to mirror the attention participants receive in the Healthy Beyond Pregnancy intervention.
  Arms: Attention Control Group

SUMMARY:
The overarching hypothesis of our research agenda is that an intervention that engages economically disadvantaged women in personalized postpartum care will promote equality in maternal child health. As a first step to test our hypothesis the investigators propose the following aims:

Specific Aim 1: Measure the impact of Healthy Beyond Pregnancy on key components of postpartum care, including use of effective contraception at three and six months postpartum and breastfeeding duration at three and six months.

Specific Aim 2: Determine if Healthy Beyond Pregnancy improves adherence to health screening and linkage to follow-up care for women with cardio-metabolic complications of pregnancy.

DETAILED DESCRIPTION:
There are profound economic inequalities in a wide range of important maternal and child health outcomes ranging from neonatal death to maternal morbidity and mortality. The overarching scientific premise for our proposal is that these inequalities stem in part from poor engagement in postpartum care by economically disadvantaged women. The investigators hypothesize that an innovative intervention grounded in empirically derived tenets of behavioral economics that includes the critical components of the American College of Obstetricians and Gynecologists (ACOG) new vision for postpartum care will narrow gaps in important maternal child health outcomes.

Women of lower socioeconomic status are at significantly increased risk of unintended pregnancies, short inter-pregnancy interval and short duration of breastfeeding. The consequences of untimed pregnancies and short duration of breastfeeding for the health of mothers, infants and children are well documented. In addition to significant health implications, these inequalities have important economic ramifications. The cost of births from unintended pregnancies in 2006 was estimated at $11 billion in maternity and infant care. This does not include cost of abortion care, lost productivity, and government assistance.

Providers have effective postpartum strategies to reduce the risk of poorly timed pregnancies and low breastfeeding rates.

Short interval or poorly timed pregnancies: Women have a range of effective contraceptive options, however, not initiating contraception postpartum remains common. The provision of long-acting reversible contraception (LARC) including intrauterine devices (IUDs) and hormonal implants has been shown to decrease short interval pregnancies and the associated risk of preterm birth. Importantly, given the array of contraceptive options available to women, it is important to make LARC accessible while empowering women to choose a method that is effective and acceptable to them. This highlights the need for solutions to engage women in patient centered comprehensive contraceptive decision-making in the postpartum period.

Short Breastfeeding Duration: A number of strategies have been shown to increase breastfeeding success. Most relevant to our proposal is that efforts to educate women about the benefits of breastfeeding, weekly text reminders in the immediate postpartum period, and access to a lactation consultant have all improved both duration and exclusivity of breastfeeding. Importantly, three recent trials demonstrated significant increases in exclusive breastfeeding from eight weeks to six months postpartum among women who received weekly-automated text message breastfeeding support. These interventions may be particularly relevant to our target population, as low-income, non-Hispanic Black women between 18-29 years send and receive text messages more frequently than any other demographic.

There are important high-risk subgroups of women who benefit uniquely from postpartum care given the need to link these women to primary or specialty health care providers in postpartum period.

Gestational diabetes (GDM): GDM complicates roughly 6-9% of pregnancies, but disproportionately burdens those with lower socio-economic status. Women with GDM are at increased risk of type 2 diabetes, metabolic syndrome, and cardiovascular disease after delivery. These findings are present as early as 3 months postpartum with the absolute risk of Type 2 diabetes approaching 5% a year postpartum. Professional societies recommend screening women for diabetes 4-12 weeks after delivery and linking women to primary care to improve long-term maternal health. In 2016, only 14% of economically disadvantaged women who received prenatal care at the Magee-Womens Hospital outpatient clinic returned for their postpartum screening. This is slightly better than national trends, which suggest roughly 6% of women with GDM had recommend postpartum screening and 13.8% had a primary care visit within a year.

Hypertensive disorders of pregnancy: Hypertensive disorders of pregnancy occur in roughly 6-8% of pregnancies and low SES is an independent risk factor. Women with hypertensive disorders of pregnancy, either gestational hypertension or preeclampsia, are more than twice as likely to develop hypertension or prehypertension in the 12 months after delivery. They are also at increased risk for cardiovascular disease. Given this, women with a hypertensive disorder of pregnancy should have early postpartum follow up for a blood pressure and establish care with a primary care physician within a year of delivery.

Recognizing the importance of the postpartum period for the health of women and children across their lifespans, ACOG recently proposed a new paradigm for postpartum care. In their new vision for postpartum care ACOG emphasized the following: 1) Postpartum care should be an on-going process rather than a single encounter 2) The content of postpartum care should be tailored to a woman's individual needs 3) The timing of the postpartum visit should be individualized for a woman. How to implement and scale this model of postpartum care and whether it will improve health outcomes for women and children has not been investigated.

Despite considerable maternal morbidity and mortality in the postpartum period, attendance rates for the postpartum visit are markedly lower for women with limited resources contributing to economic health disparities. While women with Medicaid receive excellent prenatal care, only 50% of them return for their postpartum visit. These parallel national trends, where 60% of women with Medicaid insurance return for a postpartum checkup compared with over 82% of women with private insurance. Medicaid programs serve pregnant women who are particularly vulnerable to poor health outcomes and thus this gap is critical. These data demonstrate that our current care model does not engage all women in quality postpartum care and is disproportionately failing our most vulnerable moms and babies.

Existing interventions to improve adherence with the postpartum visit have not been rigorously evaluated, would be difficult to scale, and do not reflect the new vision for postpartum care outlined by ACOG.

Empirically derived concepts from behavioral economics can be leveraged to design interventions that support patient's engagement in their health. The field of behavioral economics acknowledges that people do not make exclusively rational choices. In fact, immediate (rather than future) needs, cognitive and psychological biases, and social norms profoundly influence decision-making. Insights from the field of behavioral economics have begun to influence the health sciences as researchers seek more effective health interventions and health policy.

Healthy Beyond Pregnancy incorporates tenets of behavioral economics that address two powerful drivers of behavioral change-- awareness and willingness. Awareness has three parts: 1) an awareness of how one's behavior affects oneself 2) an awareness of how one's actions impact others and 3) an awareness of social norms around the given behavior. Awareness alone, however, is insufficient to alter behavior. People must be willing to change their behavior. Designing health interventions that address both awareness and willingness are more likely to lead to behavior change.

In the current proposal the investigators focus on four tenets of behavioral economics-bounded rationality (information overload), status quo bias (valuing the present self over the future self), hovering (limited attention), and framed incentives-- that address both awareness and willingness and have been successfully used to tackle stubborn health problems such as smoking and obesity. Both bounded rationality and hovering address awareness, while status quo bias and framed incentives address willingness.

In summary, this proposal is significant because it will evaluate the impact of an innovative program built on empirically derived concepts of behavioral economics on health decision-making in the postpartum period- a critical window for maternal child health. Our program directly mirrors the new vision for postpartum care outlined by ACOG. Additionally, it targets low-income women who are at risk for not participating in postpartum care to promote equality in maternal child health.

ELIGIBILITY:
Inclusion Criteria:

* Insured by a PA Medicaid insurance
* Pregnancy care in the Magee Womens Hospital Outpatient Clinic

Exclusion Criteria:

* Delivery less than 24 weeks
* Fetal or neonatal demise
* Women who had a postpartum tubal ligation
* Women less than 18 year of age

Ages: 12 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — This is a study of postpartum women
Enrollment: 128 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Facco, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trail will be shared immediately after publication of the trial. Data can be obtained by contacting central contact person, Katherine Himes at himekp@upmc.edu.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately upon publication of the trial. They will be available indefinitely.
Access Criteria: Anyone who wished to access the data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Attention Control Group | Pre-Scheduled Postpartum Visit: | Healthy Beyond Pregnancy
Started | 42 | 43 | 43
Completed | 42 | 43 | 43
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Attention Control Group | Pre-Scheduled Postpartum Visit: | Healthy Beyond Pregnancy | Total
Number analyzed (Participants) | 42 | 43 | 43 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (7.1) | 27 (5.2) | 27 (6.0) | 27 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 43 | 43 | 128
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 4
  Not Hispanic or Latino | 41 | 43 | 40 | 124
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 29 | 25 | 22 | 76
  White | 10 | 13 | 16 | 39
  More than one race | 3 | 4 | 4 | 11
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Using a Non-barrier Method of Contraception
Description: Effective contraception (non-barrier method)
Time Frame: 3 months after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Attention Control Group | Pre-Scheduled Postpartum Visit: | Healthy Beyond Pregnancy
Number analyzed (Participants) | 42 | 43 | 43
Participants | 24 | 29 | 22

2. Primary Outcome: Number of Participants Using a Non-barrier Method of Contraception
Description: Effective contraception (non-barrier method)
Time Frame: 6 months after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Attention Control Group | Pre-Scheduled Postpartum Visit: | Healthy Beyond Pregnancy
Number analyzed (Participants) | 42 | 43 | 43
Participants | 19 | 26 | 22

3. Primary Outcome: Adherence of Postpartum Visit
Description: Attendance at postpartum visit (yes/no)
Time Frame: 12 weeks after deliery
Measure: Count of Participants; unit: Participants
Arm/Group | Attention Control Group | Pre-Scheduled Postpartum Visit: | Healthy Beyond Pregnancy
Number analyzed (Participants) | 42 | 43 | 43
Participants | 25 | 25 | 23

4. Secondary Outcome: The Number of Participants Who Given Their Infant Breast Milk
Description: Rates of breast feeding
Time Frame: 1 week after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Attention Control Group | Pre-Scheduled Postpartum Visit: | Healthy Beyond Pregnancy
Number analyzed (Participants) | 32 | 34 | 35
Participants
  Breast Milk Only | 4 | 11 | 6
  Formula Only | 13 | 8 | 12
  Both Breast Milk and Formula | 15 | 15 | 17

5. Secondary Outcome: The Number of Participants Who Given Their Infant Breast Milk
Description: Rates of breast feeding
Time Frame: 1 month after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Attention Control Group | Pre-Scheduled Postpartum Visit: | Healthy Beyond Pregnancy
Number analyzed (Participants) | 34 | 29 | 31
Participants
  Breast Milk Only | 4 | 7 | 6
  Formula Only | 18 | 14 | 17
  Breast Milk and Formula | 12 | 8 | 8

6. Secondary Outcome: The Number of Participants Who Given Their Infant Breast Milk
Description: Rates of breast feeding
Time Frame: 3 months after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Attention Control Group | Pre-Scheduled Postpartum Visit: | Healthy Beyond Pregnancy
Number analyzed (Participants) | 23 | 25 | 26
Participants
  Breast Milk Only | 3 | 5 | 6
  Formula Only | 20 | 17 | 12
  Breast Milk and Formula | 0 | 3 | 8

7. Secondary Outcome: The Number of Participants Who Given Their Infant Breast Milk
Description: Rates of breast feeding
Time Frame: 6 months after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Attention Control Group | Pre-Scheduled Postpartum Visit: | Healthy Beyond Pregnancy
Number analyzed (Participants) | 25 | 20 | 20
Participants
  Breast Milk Only | 5 | 3 | 3
  Formula Only | 18 | 16 | 13
  Breast and Formula | 2 | 1 | 4

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Attention Control Group | Pre-Scheduled Postpartum Visit: | Healthy Beyond Pregnancy
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 0/42 | 0/43 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/52/NCT04257552/Prot_SAP_000.pdf